CLINICAL TRIAL: NCT06740227
Title: Effects of Virtual Reality-Based Balance Training Compared to Conventional Balance Training to Reduce Risk of Fall in Patients With Diabetic Peripheral Neuropathy: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/59
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Peripheral Neuropathy; Balance; Fall Risk
Keywords: Diabetic Peripheral Neuropathy (DPN); Peripheral Nervous System Disease; Hyperglycemia-Induced Neuropathy; Neuropathic Pain; Sensory Disorder; Motor Neuron Disease; Metabolic Disease; Blood Glucose Regulation Disorders; Hyperglycemia; Small Fiber Neuropathy,; Virtual Reality Based Balance Training; Conventional Balance Training; Balance Rehabilitation; Fall prevention Intervention
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia; Sensation Disorders; Motor Neuron Disease; Metabolic Diseases; Hyperglycemia; Small Fiber Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Conventional Balance Training one minute of rest for every five minutes of exercise
  Conventional Balance workout session will be for about 30-40 minutes Warm-up for 5 minutes For Static Balance, Static Balance, Single Leg Standing, Stork Standing will be used For Dynamic Balance, Weight Shifts, Tandem Walk, Single Leg Balance with Arm Movements 5 minutes will be given for cool down
  Interventions: Procedure: Conventional Balance Training
- Experimental group (Experimental): Virtual Reality based balance training
  Virtual reality workout session will be for about 30-40 minutes Warm-up exercise will be for 5 minutes including relaxed breathing For Static Balance, Lotus Focus, Tree pose, Warrior Pose games will be used For Dynamic Balance, Soccer Heading, Ski Jump, Tight Rope Walk, Table Tilt, Ski Slalom games will be used 5 minutes will be given for cool down.
  Interventions: Procedure: Virtual Reality-Based Balance Training

INTERVENTIONS:
Procedure: Virtual Reality-Based Balance Training — Virtual reality workout session will be for about 30-40 minutes Warm-up exercise will be for 5 minutes including relaxed breathing For Static Balance, Lotus Focus, Tree pose, Warrior Pose games will be used For Dynamic Balance, Soccer Heading, Ski Jump, Tight Rope Walk, Table Tilt, Ski Slalom games will be used 5 minutes will be given for cool down.
  Arms: Experimental group
Procedure: Conventional Balance Training — one minute of rest for every five minutes of exercise Conventional Balance workout session will be for about 30-40 minutes Warm-up for 5 minutes For Static Balance, Static Balance, Single Leg Standing, Stork Standing will be used For Dynamic Balance, Weight Shifts, Tandem Walk, Single Leg Balance with Arm Movements 5 minutes will be given for cool down
  Arms: Control Group

SUMMARY:
The objective of this study is to determine the effects of virtual reality based balance training compared to conventional balance training to reduce risk of fall in patients with diabetic peripheral neuropathy in terms of fall and gait parameters.

The study is a non-blinded randomized control trial, consisting of 2 groups. The Study will be conducted at Fauji Foundation Hospital and Foundation University Islamabad. A calculated sample of 30 subjects will be selected via non-probability convenience sampling technique followed by randomization into two groups using envelope method.

After CBRC registration, ethical approval is obtained from ERC FUMC. Individuals fulfilling the inclusion criteria is selected, followed by written informed consent after explaining the study purpose.

Participants is then be randomly allocated to one of the 2 groups. At the baseline, Fall Efficacy Scale (FES), Activity-specific Balance Confidence (ABC), Time Up and Go Test and Dynamic Gait Index (DGI) are assessed.

Control group is provided with conventional balance training. Treatment group is provided with the Virtual Reality (Wii Fit) Based Balance Training.

Exercise training is performed thrice a week on alternate days for a total duration of 18 sessions over 06 week.

All outcome measurements would be performed before and then after the 6-weeks intervention period.

Data will be entered and analyzed on SPSS v. 22.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 years and above
* Medical Diagnosis of diabetes under regular medication control and Diabetic Peripheral Neuropathy (DPN) confirmed
* Independent community ambulatory individuals
* Intact cognition (MMSE > 24)

Exclusion Criteria:

* Other neurological conditions I.e. Dementia, Parkinson Disease, Spinal Cord Injury or Stroke.
* Severe visual impairment, Musculoskeletal disorders, Unhealed plantar ulceration, Lower limb amputation, poor cardiopulmonary function or other disease that affects walking ability or any other disease due to which individuals are unable to walk without assistance.
* Any other condition associated with high risk of fall.
* Inability to follow simple instructions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Fear of Fall | 6 weeks
  It is a Fall Efficacy Scale (FES) is a self-revealed measure fear of fall. The FES comprises of 10 things, each addressing a typical action of day to day living, like cleaning, dressing, or walking. Respondents rate their certainty for every movement on a 10-point Likert scale, where 1 specifies "not confident at all" and 10 implies "completely confident." The all out score, got by adding the appraisals across all things, goes from 10 (least certainty) to 100 (most noteworthy certainty).
Balance | 6 weeks
  Activity Specific Balance Confidence (ABC) Scale is used particularly in assessing balance confidence among individuals, especially older adults, who may have concerns about falling during daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan